CLINICAL TRIAL: NCT01547026
Title: Self-regulation Strategies to Improve Exercise Behavior: A Randomized Clinical Trial in Persons With Schizophrenia Spectrum Disorders
Brief Title: Self-regulation Strategies to Improve Exercise Behavior Among Schizophrenic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Konstanz (Other)
Collaborators: Center for Psychiatry, Reichenau, Germany (Unknown); Thurgau Psychiatric Services, Switzerland (Unknown)
Responsible Party: Principal Investigator, Michael Odenwald, Chief Psychologist of the Schizophrenia Research Ward, University of Konstanz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UKonstanzMichaelOdenwald2012-1
Record Dates: First submitted 2012-03-03; First posted 2012-03-07 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Schizophrenia; Schizo-affective Disorder
Keywords: schizophrenia; exercise; sport; weight control; fitness
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Psycho-education (Active Comparator): Patients receive a 10 min. psycho-education on positive health effects of sports
  Interventions: Behavioral: Implementation Intentions

INTERVENTIONS:
Behavioral: Implementation Intentions — In a 10 minute structured therapy session patients are assisted to build up implementation intentions to participate in the sports program.

SUMMARY:
Patients who suffer from diseases of the schizophrenia spectrum are frequently burdened by weight gain. Sport programs have been shown to improve somatic and psychological health. However, the motivation to participate in sports therapy is usually impaired due to illness-related factors such as anhedonia and negative symptoms. Previous attempts to increase participation in sports therapy have used psycho-educational and behavioral attempts that require a lot of resources. In this study the investigators will use a brief method developed in experimental social psychology to build up implementation intentions. This method has been shown to improve psychological test performance in schizophrenia patients but has never been used in a clinical context.

In two psychiatric hospitals, in-patients with schizophrenia who have been examined by a medical doctor, for whom any medical concerns for sports therapy participation have been excluded and who declared their motivation to participate in an existing standard sports exercise program will be recruited for the study. After information on the study and signing of an informed consent patients will be randomly assigned to two treatment conditions. In the control condition, the main therapist will individually deliver a 10-minute psycho-education on the helpfulness of sports to improve the health; this will be repeated in a shorter form in the regular individual treatment sessions over the following weeks. The intervention condition will use a structured procedure of the same duration to build up implementation intentions to participate in the sports therapy. The implementation intentions will briefly be repeated and updated in the following session.

Primary outcome variables will be percentage of attended sport therapy sessions, persistence and compliance. Secondary outcome variables will be Body Mass Index. As confounding variables the investigators will assess amount of anti-psychotic medication in Chlorpromazine equivalents, negative and depressive symptoms, usual sport activities and cognitive impairments.

The investigators expect that building up implementation intentions will increase participation, persistence and compliance of the patients in the sports and exercise therapy program compared to the patients who just have received psycho-education.

ELIGIBILITY:
Inclusion Criteria:

* schizophrenia or schizo-affective disorder

Exclusion Criteria:

* manic episode
* florid positive psychotic symptoms
* catatonic symptoms
* medical concerns for possible damage to patients health by participation in sports therapy
* patient is aggressive
* patient is suicidal
* epilepsia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2012-04; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
percentage of sports therapy sessions attended | max. 8 weeks
  During a single patient's in-patient treatment, we count the number of sport therapy sessions that were attended and compute a ratio attended/offered sessions
Persistence | max. 8 weeks
  We assess whether a patient has persisted to participate in successive sports therapy session
Compliance | max. 8 weeks
  We assess how long the individual patient participates in each therapy session (standard duration 30 min.)

SECONDARY OUTCOMES:
Body Mass Index (BMI) | max. 8 weeks
  We use the routine weekly weight measurements of clinic staff to calculate changes of the BMI over the period of participation into the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Psychiatry Reichenau, Reichenau, Germany

REFERENCES:
- [Derived] Sailer P, Wieber F, Propster K, Stoewer S, Nischk D, Volk F, Odenwald M. A brief intervention to improve exercising in patients with schizophrenia: a controlled pilot study with mental contrasting and implementation intentions (MCII). BMC Psychiatry. 2015 Sep 3;15:211. doi: 10.1186/s12888-015-0513-y. PMID 26335438